CLINICAL TRIAL: NCT04366583
Title: Comparison of Hemostatic Efficacy for Argon Plasma Coagulation vs Hemoclipping Following Distilled Water Injection in Treating High-risk Bleeding Ulcers
Brief Title: Argon Plasma Coagulation vs Hemoclipping for Bleeding Peptic Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Principal Investigator, Huay-Min Wang, Division of Gastroenterology and Hepatology, Department of Internal Medicine, Kaohsiung Veterans General Hospital.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VGHKS12-CT1-17
Record Dates: First submitted 2020-04-26; First posted 2020-04-29 (Actual); Results first posted 2020-10-22 (Actual); Last update posted 2020-12-23 (Actual); Status verified 2020-11

CONDITIONS: Bleeding Peptic Ulcer
Keywords: argon plasma coagulation; hemoclipping; distilled water injection
MeSH Terms: conditions — Peptic Ulcer Hemorrhage | interventions — Argon Plasma Coagulation

STUDY DESIGN:
Intervention Model Description: Intervention device: argon plasma coagulation ( (PSD-60/Endoplasma, Olympus Corp., Tokyo,Japan) ; hemoclipping (Olympus HX 110/610) Intervention drug: distilled water design setting: argon plasma coagulation plus distilled water injection vs hemoclipping plus distilled water
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Argon plasma coagulation plus distilled water injection (Experimental): The patients in this group received Argon plasma coagulation therapy, PSD-60/Endoplasma (Olympus Corporation, Tokyo, Japan), following distilled water injection at index endoscopy. Then participants were treated with intravenous pantoprazole (Pantoloc i.v., Nycomed GmbH, Singen, Germany) 40 mg every 12 hours during the first 3 days, followed by oral pantoprazole (Pantoloc, Takeda GmbH, Oranienburg, Germany) 40 mg daily until the end of56-day study period.
  Interventions: Device: argon plasma coagulation
- Hemoclipping plus distilled water injection (Active Comparator): The patients in this group received hemoclipping (Olympus HX 110/610, Olympus Corporation, Tokyo, Japan), following distilled water injection at index endoscopy. Then participants were treated with intravenous pantoprazole (Pantoloc i.v., Nycomed GmbH, Singen, Germany) 40 mg every 12 hours during the first 3 days, followed by oral pantoprazole (Pantoloc, Takeda GmbH, Oranienburg, Germany) 40 mg daily until the end of56-day study period.
  Interventions: Device: hemoclipping

INTERVENTIONS:
Device: argon plasma coagulation — Olympus electrosurgical unit/argon plasma coagulation unit (PSD-60/Endoplasma, Olympus Corp., Tokyo, Japan)
  Arms: Argon plasma coagulation plus distilled water injection
Device: hemoclipping — clipping device (Olympus HX 110/610, Olympus Corp., Tokyo, Japan)
  Arms: Hemoclipping plus distilled water injection

SUMMARY:
Endoscopic treatment is recommended for initial hemostasis in nonvariceal upper gastrointestinal bleeding. However, the additional hemostatic efficacy of argon plasma coagulation (APC) has not been widely investigated. We designed a randomized trial comparing APC plus injection therapy vs hemoclipping plus injection therapy for peptic ulcer bleeding.

DETAILED DESCRIPTION:
【Goals and Background 】 Endoscopic treatment is recommended for initial hemostasis in nonvariceal upper gastrointestinal bleeding. Many endoscopic devices have been demonstrated to be effective in the hemostasis of bleeding ulcers. However, the additional hemostatic efficacy of argon plasma coagulation (APC) after endoscopic injection therapy has not been widely investigated.

【Study】 From Feb. 2012 to April 2016, consecutive patients with high-risk bleeding ulcers, characterized by active bleeding, non-bleeding visible vessels and adherent clots, were admitted to our hospital. They prospectively randomly underwent either APC therapy plus distilled water injection or Hemoclipping plus distilled water injection. Pantoprazole infusion was conducted during the fasting period after endoscopy and orally for 8 weeks to encourage ulcer healing. Episodes of rebleeding were retreated with endoscopic combination therapy. Patients who did not benefit from retreatment underwent emergency surgery or arterial embolization.

ELIGIBILITY:
Inclusion Criteria:

． high-risk peptic ulcer bleeding. High-risk bleeding ulcers were defined as participants with stigmata of a bleeding visible vessels (eg, spurting, oozing), a non-bleeding visible vessels (NBVV) or adherent clot.4 A NBVV at endoscopy was defined as a raised red, red-blue or pale hemispheric vessel protruding from the ulcer bed, without active bleeding. An adherent clot was defined as an overlying blood clot that was resistant to vigorous irrigation.

Exclusion Criteria:

* the presence of another possible bleeding site (eg, gastroesophageal varix, gastric cancer, reflux esophagitis)
* coexistence of actively severe ill diseases (eg, septic shock, stroke, myocardial infarction, surgical abdomen)
* treatment with an anticoagulant (eg, warfarin)
* pregnancy
* the presence of operated stomach
* refusal to participate in the study

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Actual)
Dates: Start 2012-02-09 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-04-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Wen-Chi Chen, MD, Study Director — Kaohsiung Veterans General Hospital.
Locations (1):
- Division of Gastroenterology and Hepatology, Department of Internal Medicine, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: High-risk bleeding ulcers were enrolled and defined as those with stigmata of an actively bleeding visible vessel, a non-bleeding visible vessel or adherent clots. Exclusion criteria were the presence of another possible bleeding site; coexistence of active severe illness, and systemic bleeding tendency.
Period: Overall Study
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection
Started | 82 | 84
Completed | 82 | 84
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection | Total
Number analyzed (Participants) | 82 | 84 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 25 | 45
  >=65 years | 62 | 59 | 121
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.9 (10.9) | 66.0 (12.5) | 67.0 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 22 | 53
  Male | 51 | 62 | 113
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 82 | 84 | 166
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Taiwan | 82 | 84 | 166

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Rebleeding
Description: Rebleeding was observed for a 30-day study period. One or more the following criteria were considered as evidence of recurrent bleeding: aspiration of fresh blood from a nasogastric or orogastric tube; pulse rate over 100 beats per minute; a drop in systolic blood pressure exceeding 30 mmHg; or continue coffee ground emesis or melena with a decline in hemoglobin of at least 2g/dL.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection
Number analyzed (Participants) | 82 | 84
Participants | 3 | 4

2. Secondary Outcome: Mortality
Description: all-cause deaths were recorded.
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection
Number analyzed (Participants) | 82 | 84
Participants | 0 | 1

3. Secondary Outcome: Surgery or Arterial Embolization
Description: need for surgery or arterial embolization
Time Frame: up to 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection
Number analyzed (Participants) | 82 | 84
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: 30 days
Description: Including all-cause mortality and severe adverse events (namely, procedure-induced bleeding, stricture and perforation)
Arm/Group | Argon Plasma Coagulation Plus Distilled Water Injection | Hemoclipping Plus Distilled Water Injection
All-Cause Mortality (participants affected / at risk) | 0/82 | 1/84
Serious Adverse Events (participants affected / at risk) | 1/82 | 1/84
Other Adverse Events (participants affected / at risk) | 0/82 | 0/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Argon Plasma Coagulation Plus Distilled Water Injection (N=82) | Hemoclipping Plus Distilled Water Injection (N=84)
procedure-induced bleeding (Gastrointestinal disorders) | 1 (1) | 1 (1) — the bleeding is related to a certain treatment arm
perforation (Gastrointestinal disorders) | 0 (0) | 0 (0)
stricture (Gastrointestinal disorders) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No